CLINICAL TRIAL: NCT06522737
Title: A Multicentre, Open-label, Phase 3, Randomised Controlled Trial of Duvelisib Versus Investigator's Choice of Gemcitabine or Bendamustine in Patients With Relapsed/Refractory Nodal T Cell Lymphoma With T Follicular Helper (TFH) Phenotype
Brief Title: A Study of Duvelisib Versus Gemcitabine or Bendamustine in Participants With Relapsed/Refractory Nodal T Cell Lymphoma With T Follicular Helper (TFH) Phenotype
Acronym: TERZO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBI-0145-304; 2024-516605-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma
Keywords: Nodal T Cell Lymphoma; T Follicular Helper; Relapsed/Refractory; Duvelisib; Peripheral T cell lymphoma; Angioimmunoblastic T cell lymphoma; TERZO; 145-304; TFH
MeSH Terms: conditions — Lymphoma; Recurrence; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy | interventions — duvelisib; Gemcitabine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duvelisib (Experimental): Duvelisib will be administered orally twice daily (BID) in 28-day cycles.
  Interventions: Drug: Duvelisib
- Gemcitabine or Bendamustine (Active Comparator): Participants will receive the investigator's choice of gemcitabine or bendamustine. The regimen to be used after randomization must be selected by the investigator prior to randomization. Gemcitabine will be administered intravenously (IV) on days 1, 8, and 15 of each 28-day cycle for up to 6 cycles. Bendamustine will be administered IV on days 1 and 2 of each 21-day cycle for up to 6 cycles.
  Interventions: Drug: Gemcitabine; Drug: Bendamustine

INTERVENTIONS:
Drug: Duvelisib — oral capsules
  Arms: Duvelisib
Drug: Gemcitabine — solution for intravenous infusion
  Arms: Gemcitabine or Bendamustine
Drug: Bendamustine — solution for intravenous infusion
  Arms: Gemcitabine or Bendamustine

SUMMARY:
The study will evaluate the progression-free survival benefit of duvelisib monotherapy as compared to investigator's choice of gemcitabine or bendamustine in participants with relapsed/refractory nodal T cell lymphoma with TFH phenotype.

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically confirmed nodal T cell lymphoma with TFH phenotype according to the criteria of the World Health Organization classification (Swerdlow 2017, Alaggio 2022) including any one of Angioimmunoblastic T cell lymphoma (AITL), follicular T cell lymphoma, and other nodal peripheral T cell lymphoma (PTCL) with a TFH phenotype.
* Relapsed or refractory to at least 1 prior systemic, cytotoxic therapy for T cell lymphoma.
* Measurable disease as defined by Lugano 2014 criteria (Cheson 2014) for T cell lymphoma.

Key Exclusion Criteria:

* Cutaneous-only disease.
* Received prior allogeneic transplant any time in the past or received autologous transplant within 60 days prior to the first dose of study drug.
* Received prior treatment with a phosphoinositide-3-kinase (PI3K) inhibitor.
* Prior exposure to planned study treatment investigator's choice therapy (gemcitabine or bendamustine) within 60 days prior to the first dose of study drug.

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as assessed by the Independent Review Committee (IRC) | Up to 3 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years
PFS as assessed by the investigator | Up to 3 years
Objective Response Rate (ORR) as assessed by the IRC | Up to 3 years
Complete Response Rate (CRR) as assessed by the IRC | Up to 3 years
Duration of Response (DOR) as assessed by the IRC | Up to 3 years
Proportion of participants who proceed to Stem Cell Transplantation (SCT) | Up to 3 years
Investigator-assessed PFS in participants who proceed to SCT | Up to 3 years
Number of participants with Adverse Events (AEs) | Up to 3 years
Quality of Life (QoL): European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Score | Up to 3 years
QoL: EQ5D Score | Up to 3 years
QoL: QLQ-NHL-HG29 Score | Up to 3 years
Concentration of Duvelisib and its Metabolites in Blood | Day 1 of Cycle 1 and Cycle 2 (predose and 60 minutes postdose)

CONTACTS AND LOCATIONS:
Locations (43):
- Belgium (2):
  - Universitair Ziekenhuis Gent (UZ Gent), Ghent
  - UZ Leuven - Gasthuisberg Campus, Leuven
- Vseobecna fakultni nemocnice, Prague, Czechia
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
  - Odense Hospital, Odense
- France (11):
  - UNICANCER - Centre Henri-Becquerel, Rouen, Normandy
  - Institut Gustave Roussy, Villejuif, Vaillant
  - CHU Cote de Nacre, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hopital Pitie Salpetriere, Paris
  - CHU Bordeaux, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU PONTCHAILLOU-Haematology, Rennes
  - Institut Curie Paris, Saint-Cloud
- Germany (4):
  - Evangelisches Krankenhaus Essen-Werden, Essen
  - Universitaetsmedizin Goettingen (UMG) - Klinik fuer Haematologie und Medizinische Onkologie, Goettigen
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaetsklinikum Leipzig- Klinik und Poliklinik fuer Haematologie und Zelltherapie, Leipzig
- Italy (5):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo - Alessandria, Alessandria
  - Asst Papa Giovanni Xxiii Uo Ematologia, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Ematologia Oncologia Instituto Pascale, Naples
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Netherlands (2):
  - Amsterdam UMC location AMC, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne Oddzial Hematologii i Transplantologii, Gdansk
  - Pratia Centrum Medyczne Krakow, Krakow
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej - Curie, Warsaw
- Spain (4):
  - ICO Hospitalet (Hospital Duran i Reynals), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (7):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - UCLH NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No